CLINICAL TRIAL: NCT03562169
Title: A Phase III Study to Determine the Role of Ixazomib as an Augmented Conditioning Therapy in Salvage Autologous Stem Cell Transplant (ASCT) and as a Post-ASCT Consolidation and Maintenance Strategy in Patients With Relapsed Multiple Myeloma
Brief Title: The Role of Ixazomib in Autologous Stem Cell Transplant in Relapsed Myeloma - Myeloma XII (ACCoRd)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Cancer Research UK (Other); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM16/047; 2016-000905-35 (EudraCT Number)
Record Dates: First submitted 2016-12-06; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Autologous Stem Cell Transplant (ASCT) (Active Comparator): Melphalan 200mg/m2 IV infusion on Day -1, followed by ASCT on Day 0
  Interventions: Drug: Ixazomib, thalidomide, & dexamethasone (ITD) re-induction; Drug: Conventional autologous stem cell transplant (ASCT-con); Drug: ITD consolidation and ixazomib maintenance vs. No further therapy
- Augmented Autologous Stem Cell Transplant (ASCT) (Experimental): Melphalan 100mg/m2 IV infusion on Day -3 and -2 plus ixazomib 4mg capsules on Day -4 and -1. ASCT will then be given on Day 0.
  Interventions: Drug: Ixazomib, thalidomide, & dexamethasone (ITD) re-induction; Drug: Augmented autologous stem cell transplant (ASCT-aug); Drug: ITD consolidation and ixazomib maintenance vs. No further therapy

INTERVENTIONS:
Drug: Ixazomib, thalidomide, & dexamethasone (ITD) re-induction — 4 - 6 ITD 28-day cycles as follows:
  * Ixazomib 4mg capsule on days 1, 8 and 15
  * Thalidomide 100mg capsule on days 1-28
  * Dexamethasone 40mg tablets on days 1, 8, 15 and 22
Drug: Conventional autologous stem cell transplant (ASCT-con) — Melphalan 200mg/m2 IV infusion on Day -1, followed by ASCT on Day 0.
  Arms: Conventional Autologous Stem Cell Transplant (ASCT)
Drug: Augmented autologous stem cell transplant (ASCT-aug) — Melphalan 100mg/m2 IV infusion on Day -3 and Day -2 plus ixazomib 4mg capsules on Day -4 and Day -1. ASCT will then be given on Day 0.
  Arms: Augmented Autologous Stem Cell Transplant (ASCT)
Drug: ITD consolidation and ixazomib maintenance vs. No further therapy — Participants will be randomised to either 'no further therapy' or 'ITD consolidation and ixazomib maintenance'. Participants randomised to 'no further treatment' will not receive any further treatment but will be followed up at 8 weeks post randomisation 2 and at 3-monthly clinic visits until disease progression.
  Participants randomised to ITD consolidation and ixazomib maintenance will receive:
  Two 28-day cycles of ITD consolidation (same doses as in ITD re-induction). This will be followed by ixazomib maintenance as follows: Ixazomib 4mg capsule on days 1, 8 and 15 of each 28-day cycle until disease progression.

SUMMARY:
Study design: Randomised, controlled, multi-centre, open-label, phase III trial (with a single intervention registration phase).

Primary Objectives

The primary objectives of this study are to determine:

* The impact on Depth of Response (DoR: less than VGPR versus VGPR or better) when salvage ASCT conditioning is augmented by the addition of a proteasome inhibitor
* The influence of a consolidation and maintenance strategy on the Durability of Response (DuR:PFS)

Secondary objectives

The secondary objectives of this study are to determine:

* Overall survival
* Time to disease progression
* The overall response rate following ixazomib, thalidomide and dexamethasone (ITD) re-induction
* Time to next treatment
* Progression-free survival 2 (PFS2)
* Duration of response
* Minimal Residual Disease (MRD) negative rate post re-induction, post-ASCT and conversion after ITD consolidation
* Engraftment kinetics
* Toxicity and safety
* Quality of life (QoL)

Participant population (refer to protocol section 9 for a full list of eligibility criteria).

* Relapsed MM (with measurable disease by IMWG criteria) previously treated with ASCT
* First progressive disease (PD) at least 12 months since first ASCT, requiring therapy.
* ECOG Performance Status 0-2
* Aged at least 18 years
* Adequate full blood count and renal, hepatobiliary, pulmonary and cardiac function
* Written informed consent

Interventions: All participants will be registered at trial entry and will receive re-induction therapy with 4-6, 28-day cycles of ixazomib, thalidomide and dexamethasone (ITD), in order to reach maximum response. Participants who achieve at least stable disease (SD) will be randomised on a 1:1 basis to receive either conventional ASCT (ASCTCon), using melphalan, or augmented ASCT (ASCTAug), using melphalan with ixazomib. All participants achieving or maintaining a minimal response (MR) or better following trial ASCT will undergo a second randomisation to consolidation and maintenance or no further treatment. Participants randomised to consolidation and maintenance will receive treatment as follows: consolidation with 2 cycles of ITD and maintenance with ixazomib until disease progression.

Number of participants: 406 participants will be registered into the trial to allow 284 participants to be randomised at the first randomisation (R1) and 248 participants to be randomised at the second randomisation (R2).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with relapsed MM (with measurable disease, according to IMWG criteria (Appendix 2)) previously treated with ASCT).
2. First Progressive Disease (PD) at least 12 months following first ASCT, requiring therapy.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 (Appendix 3).
4. Aged at least 18 years.
5. Participants must have the following blood results within 14 days before registration:

   1. Absolute neutrophil count (ANC) ≥1x109/L
   2. Platelet count ≥75x109/L. If the participant has ≥50% bone marrow infiltration a platelet count of ≥50x109/L is allowed.

   Platelet transfusions are not allowed within 3 days before registration in order to meet these values.
6. Adequate renal function within 14 days before registration:

   a. Creatinine clearance ≥30ml/min (calculated according to the Cockcroft-Gault equation or other locally approved formula)
7. Adequate hepatobiliary function within 14 days before registration:

   1. Total bilirubin <2 x upper limit of normal (ULN)
   2. ALT <2 x ULN
8. Adequate pulmonary function within 14 days before registration:

   a. Adequate respiratory functional reserve (delineated by KCO/DLCO (carbon monoxide diffusion in the lung) of ≥50%). No evidence of a history of pulmonary disease. If a significant history, then a review by a respiratory medicine physician is required.
9. Adequate cardiac function within 12 weeks before registration

   a. Left ventricular ejection fraction (LVEF) ≥40%. Note: repeat confirmation of cardiac function is needed if treatment is given between this assessment and registration.
10. Female participants who:

    1. Are not of childbearing potential (Appendix 8), OR
    2. If they are of childbearing potential (Appendix 8), agree to practice 2 effective methods of contraception (Appendix 8), at the same time, from the time of signing the informed consent form until 90 days after the last dose of study drug, OR
    3. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

    Male participants, even if surgically sterilised (i.e. status post-vasectomy), must agree to one of the following:
    1. Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
    2. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.) Contraception for female and male participants must be in accordance with (and consent to) the Celgene-approved Thalidomide Pregnancy Prevention Programme.
11. If female and of childbearing potential (see Appendix 8), must have a negative pregnancy test performed by a healthcare professional in accordance with the Celgene Thalidomide Pregnancy Prevention Programme.
12. Patients agree not to receive other clinical trials treatment, including investigational medicinal products (IMPs) not included in this trial, within 30 days of trial registration and throughout the duration of the trial, until disease progression.
13. Able to provide written informed consent.

Exclusion Criteria:

1. Received prior second line therapy for their relapsed disease other than local radiotherapy, therapeutic plasma exchange, or dexamethasone (up to a maximum of 200mg is allowed but not within 30 days prior to registration). Radiotherapy sufficient to alleviate or control pain of local invasion is permitted, but must not be within 14 days before registration. Patients who have received hemi-body radiation or similar since relapse will not be eligible.
2. ≥Grade 2 peripheral neuropathy within 14 days before registration.
3. Known HIV seropositivity.
4. Known resistance, intolerance or sensitivity to any component of the planned therapies.
5. Any medical or psychiatric condition which, in the opinion of the investigator, contraindicates the participant's participation in this study.
6. Previous or concurrent malignancies at other sites (excluding completely resected non-melanoma skin cancer or carcinoma in situ of any type, such as cervical cancer).
7. Pregnant, lactating or breast feeding female participants.
8. Failure to have fully recovered (i.e.Grade 1 or less toxicity) from the reversible effects of prior chemotherapy.
9. Major surgery within 14 days before registration.
10. Central nervous system involvement with myeloma.
11. Ongoing or active infection requiring systemic antibiotic therapy or other serious infection within 14 days before registration.
12. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
13. Systemic treatment, within 14 days before the first dose of ixazomib with strong CYP3A inducers (e.g. rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
14. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib, including difficulty swallowing.
15. Patients that have previously been treated with ixazomib or participated in a study with ixazomib whether treated with ixazomib or not.
16. Participant has current or prior hepatitis B or C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 100 days post-ASCT
  Overall response rate following ASCT will be determined according to the IMWG Uniform Response Criteria for Multiple Myeloma. This endpoint will be defined as a binary dichotomization of response (≥VGPR vs <VGPR) at an assessment 100 days after the date of stem cell transplant.
Progression-free survival | From date of registration to date of disease progression, up to 120 months.
  The influence of a consolidation and maintenance strategy on the Durability of Response (DuR: PFS)

SECONDARY OUTCOMES:
Overall survival | From date of R2 to date of death, up to 120 months
  Overall survival is defined as the time from randomisation to the consolidation/maintenance part of the trial post-ASCT to death from any cause or last follow-up.
Time to disease progression | From date of registration until date of disease progression, up to 120 months
  Time to disease progression is defined as time from randomisation to the consolidation/maintenance part of the trial post-ASCT to first documented evidence of disease progression. Participants who die without disease progression will be censored in the analysis.
Overall response rate to ITD re-induction | At the end of re-induction - after 4-6 re-induction cycles (each cycle is 28 days)
  Overall response rate following re-induction will be determined according to the IMWG Uniform Response Criteria for Multiple Myeloma.
Upgrade in response after two cycles of ITD consolidation | After 2 cycles of ITD consolidation (each cycle is 28 days)
  Upgrade in response after 2 cycles of ITD consolidation - response rate following ITD consolidation will be determined according to the IMWG Uniform Response Criteria for Multiple Myeloma. This endpoint will be defined as a binary dichotomization of response (≥VGPR vs <VGPR).
Progression-free survival 2 (PFS2) | Date of R2 to date of second disease progression, up to 120 months
  Progression-free survival 2 is defined as the time from second randomisation to the consolidation/maintenance part of the trial post-ASCT to second documented disease progression (or the start of next line anti-myeloma treatment), or death from any cause, whichever occurs first. Participants alive and for whom a second progression after second randomisation has not been observed will be censored at the last day they were known to be alive and second progression-free.
Time to next treatment | Date of registration to start date of new therapy, up to 120 months
  Time to next line treatment is defined as the time from the date of randomisation to the date of commencement of next line treatment. Participants who do not receive next line treatment will be censored at the date of the last assessment or follow-up visit where they are known to have received no new therapy.
Duration of response | Date of achieving at least partial response to date of disease progression, up to 120 months
  Duration of response to protocol treatment is defined from the time of achieving at least a partial response to the date of first documented evidence of disease progression. Participants who die prior to documentation of disease progression will be censored at the date of death. Participants dying from causes not primarily due to progression will also be censored at the date of death. Participants not reaching disease progression at the time of analysis will be censored at the last date known to be progression-free.
Proportion of patients Minimal Residual Disease negative | Baseline; End of re-induction (after 4-6 cycles of re-induction, each cycle is 28 days); 100 days post-ASCT; After 2 cycles of consolidation (each cycle is 28 days); 8 weeks post-randomisation 2; 12 months post-randomisation 2
  Proportion of patients Minimal Residual Disease negative is defined as the proportion of participants with minimal residual disease (MRD) negative as assessed by flow cytometry will be assessed at various points in trial protocol treatment.
Continuous Minimal Residual Disease (MRD) | Baseline; End of re-induction (after 4-6 cycles of re-induction, each cycle is 28 days); 100 days post-ASCT; After 2 cycles of consolidation (each cycle is 28 days); 8 weeks post-randomisation 2; 12 months post-randomisation 2
  Continuous Minimal Residual Disease (MRD) measurements as assessed by flow cytometry will be assessed at various points in trial protocol treatment.
Engraftment kinetics_test | Stem cell harvest; 100 days post-ASCT
  Engraftment kinetics will be summarised based on summaries of stem cell remobilisation protocol and success of remobilisation and stem cell harvest after the completion of ASCT for all participants.
Incidence of treatment-emergent adverse events (Toxicity and safety) | Baseline; End of each re-induction cycle (each cycle is 28 days); 100 days post-ASCT; End of 2 cycles of consolidation (each cycle is 28 days); 8 weeks post-R2; 3 monthly post-R2 until disease progression; Disease progression, up to 120 months
  Toxicity and safety will be reported based on adverse events, as graded by CTCAE V4.03 and determined by routine clinical assessments at each centre.
EORTC QLQ-C30_questionnaire | Baseline; End of re-induction (after 4-6 cycles of re-induction, each cycle is 28 days); 100 days post-ASCT; 12 months post-R2; 24 months post-R2
  The EORTC QLQ-C30 questionnaire will be used to measure participant-assessed quality of life at registration, post re-induction, 100 days post-ASCT and annually post second randomisation until 24 months post second randomisation, or until disease progression whichever is earlier.
EORTC QLQ-MY20_questionnaire | Baseline; End of re-induction (after 4-6 cycles of re-induction, each cycle is 28 days); 100 days post-ASCT; 12 months post-R2; 24 months post-R2
  The EORTC QLQ-MY20 questionnaire will be used to measure participant-assessed quality of life at registration, post re-induction, 100 days post-ASCT and annually post second randomisation until 24 months post second randomisation, or until disease progression whichever is earlier.
EQ-5D_questionnaire | Baseline; End of re-induction (after 4-6 cycles of re-induction, each cycle is 28 days); 100 days post-ASCT; 12 months post-R2; 24 months post-R2
  The EQ-5D questionnaire will be used to measure participant-assessed quality of life at registration, post re-induction, 100 days post-ASCT and annually post second randomisation until 24 months post second randomisation, or until disease progression whichever is earlier.

OTHER OUTCOMES:
Cytogenetics_composite measure | Through study completion, up to 120 months
  Cytogenetic subgroups will be analysed to explore a number of specific hypotheses, including the effect on PFS, OS, TTP and response (≥VGPR vs. <VGPR). Some examples of what will be studied include chromosome 14 translocations and abnormalities of chromosome 1p, 1q, 13q and 17p. In addition, other regions considered to be of interest will be analysed according to the statistical analysis plan. Other subgroup and exploratory analyses may also be carried out and will be described in the statistical analysis plan or separate analyses plans related to translational work.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Trial Management, Study Director — Univeristy of Leeds, CTRU
Locations (91):
- United Kingdom (91):
  - Aberdeen Royal Infirmary, Aberdeen
  - Monklands Hospital, Airdrie
  - University Hospital Ayr, Ayr
  - Barnsley Hospital, Barnsley
  - Basingstoke & North Hampshire Hospital, Basingstoke
  - Royal United Hospital, Bath
  - Good Hope Hospital, Birmingham
  - Heartlands Hospital, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Pilgrim Hospital, Boston
  - Royal Bournemouth Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Bristol Haematology & Oncology Centre, Bristol
  - Southmead Hospital, Bristol
  - Queen's Hospital, Burton-on-Trent
  - Addenbrooke's Hospital, Cambridge
  - St Helier Hospital, Carshalton
  - Cheltenham General Hospial, Cheltenham
  - Countess of Chester Hospital, Chester
  - Chesterfield Royal Hospital, Chesterfield
  - St Richards Hospital, Chichester
  - University Hospital Coventry, Coventry
  - Royal Derby Hospital, Derby
  - Dewsbury Hospital, Dewsbury
  - Russells Hall Hospital, Dudley
  - Ninewells Hospital, Dundee
  - Hairmyres Hospital, East Kilbride
  - Western General Hospital, Edinburgh
  - Beatson Cancer Centre, Glasgow
  - New Victoria Hospital, Glasgow
  - Gloucestershire Royal Hospital, Gloucester
  - Grantham and District Hospital, Grantham
  - Diana Princess of Wales Hospital, Grimsby
  - Calderdale Royal Hospital, Halifax
  - Harrogate District Hospital, Harrogate
  - Huddersfield Royal Infirmary, Huddersfield
  - Castle Hill Hospital, Hull
  - Raigmore Hospital, Inverness
  - Ipswich Hospital, Ipswich
  - Kidderminster Hospital, Kidderminster
  - University Hospital Crosshouse, Kilmarnock
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - Royal Liverpool University Hospital, Liverpool
  - University Hospital Aintree, Liverpool
  - Guys and St Thomas's Hospital, London
  - Kings College Hospital, London
  - Royal Marsden Hospital, London
  - St Barts Hospital, London
  - University College London Hospital, London
  - Maidstone Hospital, Maidstone
  - Manchester Royal Infirmary, Manchester
  - The Christie, Manchester
  - Borders General Hospital, Melrose
  - James Cook University Hospital, Middlesbrough
  - Milton Keynes General Hospital, Milton Keynes
  - Freeman Hospital, Newcastle
  - North Tyneside General Hospital, North Shields
  - Norfolk & Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Royal Oldham Hospital, Oldham
  - Churchill Hospital, Oxford
  - Royal Alexandra Hospital, Paisley
  - Derriford Hospital, Plymouth
  - Pontefract Hospital, Pontefract
  - Whiston Hospital, Prescot
  - Royal Berkshire Hospital, Reading
  - Redditch Hospital, Redditch
  - Tunbridge Wells Hospital, Royal Tunbridge Wells
  - Salford Royal Hospital, Salford
  - Salisbury Hospital, Salisbury
  - Scunthorpe General Hospital, Scunthorpe
  - Royal Hallamshire Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - St Helens Hospital, St Helens
  - Stafford County Hospital, Stafford
  - Stepping Hill Hospital, Stockport
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - King's Mill Hospital, Sutton in Ashfield
  - Singleton Hospital, Swansea
  - Musgrove Park Hospital, Taunton
  - St George's Hospital, Tooting
  - Pinderfields General Hospital, Wakefield
  - Royal Hampshire County Hospital, Winchester
  - Wishaw Hospital, Wishaw
  - New Cross Hospital, Wolverhampton
  - Worcestershire Royal Hospital, Worcester
  - Worthing Hospital, Worthing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Striha A, Ashcroft AJ, Hockaday A, Cairns DA, Boardman K, Jacques G, Williams C, Snowden JA, Garg M, Cavenagh J, Yong K, Drayson MT, Owen R, Cook M, Cook G. The role of ixazomib as an augmented conditioning therapy in salvage autologous stem cell transplant (ASCT) and as a post-ASCT consolidation and maintenance strategy in patients with relapsed multiple myeloma (ACCoRd [UK-MRA Myeloma XII] trial): study protocol for a Phase III randomised controlled trial. Trials. 2018 Mar 7;19(1):169. doi: 10.1186/s13063-018-2524-8. PMID 29514706
- See also: Myeloma XII protocol paper — https://www.ncbi.nlm.nih.gov/pubmed/29514706